CLINICAL TRIAL: NCT01291420
Title: Therapeutic Efficacy of Wilms' Tumor Gene (WT1) MRNA-electroporated Autologous Dendritic Cell Vaccination in Patients with Solid Tumors: a Phase I/feasibility Study
Brief Title: Dendritic Cell Vaccination for Patients with Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Zwi Berneman, MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG 11-001
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma; Renal Cell Carcinoma; Sarcomas; Breast Cancers; Malignant Mesothelioma; Colorectal Tumors
MeSH Terms: conditions — Glioblastoma; Carcinoma, Renal Cell; Sarcoma; Breast Neoplasms; Mesothelioma, Malignant; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: autologous dendritic cell vaccination — 4 biweekly intradermal DC injections of 10*10E6 DCs (500 µL) at 5 sites (100 µL/site) in the ventromedial regions of the upper arm approximately 5-10 cm of the regional lymph nodes

SUMMARY:
The aim of this study is to evaluate the immunogenicity and clinical efficacy of intradermal vaccination with autologous RNA-modified dendritic cells (DCs) - engineered to express the WT1 protein - in patients with limited spread metastatic solid tumors, i.e. breast cancers, glioblastoma grade IV, sarcomas, malignant mesothelioma and colorectal tumors. Based on the results of our previously performed phase I study with autologous WT1 mRNA-transfected DC, the investigators hypothesize that the vaccination with DC will be well-tolerated and will result in an increase in WT1-specific CD8+ T cell responses.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor type:

   Metastatic or Locally Advanced Breast Cancer; Malignant Mesothelioma; Glioblastoma Multiforme (Grade IV); Sarcoma's; Colorectal tumors or rare tumors (less than 500 patients a year)
2. Extent of disease:

   * Metastatic Breast Cancer or High Risk Locally Advanced Breast Cancer

     * Partial or Complete response after first line chemotherapy for both metastatic or locally advanced breast cancer. Minimal metastatic disease under hormonal treatment
     * High risk Locally Advanced breast cancer defined as (and/or):

       * Age < 60 years old
       * ER, PR and Her-2 Neu negative tumors
       * > 4 lymphnodes at initial presentation
       * Mastitis Carcinomatosis
       * Pregnancy associated Breast Cancer
   * Malignant Mesothelioma:

     * Partial or Complete response after first line chemotherapy not amendable for surgery
     * Adjuvant after debulking surgery
   * Glioblastoma Multiforme

     * In Recurrent Disease after optimal treatment according to Stupp regimen
     * In primary disease after debulking surgery, Temodal/radiotherapy and Temodal chemotherapy for 6 months
   * Sarcoma's

     * After adjuvant chemotherapy for uterine sarcoma's
     * After Optimal or Debulking Surgery for liposarcoma's, synovial cell sarcoma's
     * Recurrent sarcoma's with limited disease
   * Colorectal tumors

     * K-ras wild-type tumors with inoperable lymphnode metastasis after standard chemotherapy (FOLFOX, FOLFIRI)
3. Patient Characteristics

   * Prior treatments: Patients must have received at least one prior chemotherapeutic regimen and must be more than 1 month past the last treatment.
   * Age: ≥ 18 years old
   * Performance status: WHO PS grade 0-1 (Appendix B)
   * Objectively assessable parameters of life expectancy: more than 3 months
   * Prior and concomitant associated diseases allowed with the exception of underlying autoimmune disease and positive serology for HIV/HBV/HCV
   * No concomitant use of immunosuppressive drugs, hormonal treatment for breast cancer is allowed in case of stable disease
   * Adequate renal and liver function, i.e. creatinin and bilirubin = 1.2 times the upper limit of normal
   * Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
   * Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

1. Subjects with concurrent additional malignancy (with exception of non-melanoma skin cancers and carcinoma in situ of the cervix)
2. Subjects who are pregnant
3. Subjects who have sensitivity to drugs that provide local anesthesia
4. Subjects needing corticosteroids 1 mg/kg during vaccination; corticosteroids are allowed as part of their treatment when taken ≥ 30 days before the start of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of intradermal DC vaccination | up to 2 months
  Immunogenicity of intradermal DC vaccination (cellular + humoral immunity against WT1 antigen) as measured by:
  1. In vivo cytokine response (serum concentration of cytokines)
  2. In vivo anti-WT1 antibody responses
  3. In vitro T cell reactivity towards MHC class I and II-restricted WT1 epitopes by multiplex-cytokine assay using peripheral blood and DTH-infiltrating T cells
  4. Delayed type hypersensitivity (DTH) responses
  5. Quantitative and qualitative FACS analysis of WT1-specific-positive CD8+ T cells using HLA-A2 WT1 multimers

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Center for Cellular Therapy and Regenerative Medicine, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Background] Van Driessche A, Van de Velde AL, Nijs G, Braeckman T, Stein B, De Vries JM, Berneman ZN, Van Tendeloo VF. Clinical-grade manufacturing of autologous mature mRNA-electroporated dendritic cells and safety testing in acute myeloid leukemia patients in a phase I dose-escalation clinical trial. Cytotherapy. 2009;11(5):653-68. doi: 10.1080/14653240902960411. PMID 19530029